CLINICAL TRIAL: NCT06292429
Title: Effects of Complex Training on Physical Fitness, Bowling Performance, Work Capacity, Muscle Strength and Bone Density in Cricket Fast Bowlers
Brief Title: Effects of Complex Training in Cricket Fast Bowlers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/1104
Record Dates: First submitted 2024-01-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Resistance Training; Plyometric Exercise; Sports Physical Therapy
Keywords: Complex Training; Cricket Fast Bowlers
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complex Training (Experimental)
  Interventions: Other: Complex Training
- Conventional Training (Active Comparator)
  Interventions: Other: Conventional Training
- Control Group (Other)
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Complex Training — Week 1-4: Foundation Phase Lower Body Resistance Training Squats (Back Squats or Goblet Squats) Deadlifts Lunges
  Paired with:
  Box Jumps Depth Jumps
  Upper Body Resistance Training Bench Press Overhead Press
  Paired with:
  Medicine Ball Chest Pass Medicine Ball Overhead Throw Rows (Barbell or Dumbbell)
  Week 5-8: Strength and Power Phase Lower Body Resistance Training Power Cleans Front Squats Romanian Deadlifts
  Paired with:
  Box Jumps with Barbell Depth Jumps with Medicine Ball
  Upper Body Resistance Training Push Press Pull-Ups or Lat Pulldowns Bent Over Rows
  Paired with:
  Plyometric Push-Ups Medicine Ball Slam
  Week 9-12: Power and Speed Phase Lower Body Resistance Training Snatch Split Squats Jumping Lunges
  Paired with:
  Box Jumps with Barbell Depth Jumps with Medicine Ball
  Upper Body Resistance Training Speed Bench Press Face Pulls Plyometric Pull-Ups
  Paired with:
  Medicine Ball Chest Pass Medicine Ball Overhead Throw
  Arms: Complex Training
Other: Conventional Training — Week 0-4 Session 1 Rotator cuff wall compression Forearm flexor compression Alpha ball tricep scrape Band assisted pushups Session 2 Soft ball thoracic breathing Neck ball arm rotations ITb compressions Middle quard compressions
  Week 4-8 Session 1 Kneeling pall of band hold Kneeling pall of partner proturbations Leg lower with mediball neutral Half lying arm speed and swing drill Session 2 Single leg band hold Trunk activated psoas lowers Split clam Bulgarian split iso hold
  Week 8-12 Session 1 Point kneel thoracic rotations Side lying single arm thoracic abduction Banded side lying clams Side lying abduction from glute Session 2 Low back mobility Kneeling pall off band hold Clean and jerks power drill movements Weighted bench press Session 3 Standing band rotations thoracic only Band pull aparts Tennis ball in trap arm flexion ext thumb to floor Bulgarian weighted
  Arms: Conventional Training
Other: Control Group — No intervention given
  Arms: Control Group

SUMMARY:
This study will be a randomized controlled trial and the data will be collected from National Cricket Academy and domestic cricket clubs. The sample size will be calculated by conducting a pilot study. There will be three groups. Group-A will be receiving Complex training, Group-B will be receiving Conventional training and Group C as a Control Group. Athletes with same physical fitness level will be recruited. There will be parallel assignment of the participants. Assessor will be kept blinded. All the parameters would be assessed at Baseline, 6 Weeks, 12 Weeks. Physical fitness will be assessed through Field Testing. Bowling performance will be assessed through speed machine and Kinovea Software. Work capacity will be assessed through step testing. Muscle strength will be assessed through Dynamometer. Lastly, BMD will be assessed though Bone Densitometer.

DETAILED DESCRIPTION:
Cricket fast bowlers require a unique blend of speed, strength, power, and agility to excel in their role on the field. In recent years, Complex training has emerged as a popular training method to enhance these critical qualities among fast bowlers. Complex training involves combining strength exercises with explosive, sport-specific movements in a single training session, aiming to improve overall athletic performance. This study will be a randomized controlled trial and the data will be collected from National Cricket Academy and domestic cricket clubs. The sample size will be calculated by conducting a pilot study. There will be three groups. Group-A will be receiving Complex training, Group-B will be receiving Conventional training and Group C as a Control Group. Athletes with same physical fitness level will be recruited. There will be parallel assignment of the participants. Assessor will be kept blinded. All the parameters would be assessed at Baseline, 6 Weeks, 12 Weeks. Physical fitness will be assessed through Field Testing. Bowling performance will be assessed through speed machine and Kinovea Software. Work capacity will be assessed through step testing. Muscle strength will be assessed through Dynamometer. Lastly, BMD will be assessed though Bone Densitometer.

ELIGIBILITY:
Inclusion Criteria:

* Male bowlers between 18 - 25 years
* Bowling speed 115-130 km/h
* Same Run-up speed (20-25 km/h)
* domestic teams
* Active in game from last 6 months
* Athletes with same 1 Repetition Maximum (Bench press and Leg press)
* Athletes with same BMI category (18.5 - 24.9)

Exclusion Criteria:

* Red flags
* Resistance training from last 6 months
* Any disabling musculoskeletal injury
* Glenohumeral Internal Rotation Deficit
* Scapular Dyskinesia
* Athletes taking prohibited drugs, Ergogenic aids
* Any cardiovascular issue . Any systemic disease

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Physical fitness (linear speed capability) | 0 week, 6 week, 12 week
  will be assessed by lower body vertical jump test
Physical fitness (lower limb explosive power) | 0 week, 6 week, 12 week
  will be assessed by 20-m sprint test
Physical fitness (upper body strength test) | 0 week, 6 week, 12 week
  will be assessed by bench press & bent over row
Physical fitness (lower body strength test) | 0 week, 6 week, 12 week
  will be assessed by hex-bar deadlift
Physical fitness (upper body muscular endurance) | 0 week, 6 week, 12 week
  will be assessed by horizontal pull
Physical fitness (aerobic capacity) | 0 week, 6 week, 12 week
  will be assessed by Yo-Yo intermittent recovery Level 1 test
Bowling performance (Ball speed) | 0 week, 6 week, 12 week
  will be measured by Pocket Radar
Bowling performance (run-up time) | 0 week, 6 week, 12 week
  will be measured by Dartfish software
Bowling performance (accuracy) | 0 week, 6 week, 12 week
  will be measured by Dartfish software
Bowling performance (RPE) | 0 week, 6 week, 12 week
  will be measured by Borg scale

SECONDARY OUTCOMES:
Work capacity | 0 week, 6 week, 12 week
  will be assessed by Step Testing
Muscle Strength | 0 week, 6 week, 12 week
  will be assessed by Hand-held Dynamometer
Bone Density | 0 week, 6 week, 12 week
  will be assessed by Bone Densitometer

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Atif Javed, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board Coaching Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feros SA, Young WB, O'Brien BJ. Efficacy of Combined General, Special, and Specific Resistance Training on Pace Bowling Skill in Club-Standard Cricketers. J Strength Cond Res. 2020 Sep;34(9):2596-2607. doi: 10.1519/JSC.0000000000002940. PMID 30741863
- [Background] Harrison DC, Doma K, Leicht AS, McGuckin TA, Woods CT, Connor JD. Repeated Bout Effect of Two Resistance Training Bouts on Bowling-Specific Performance in Male Cricketers. Sports (Basel). 2022 Aug 24;10(9):126. doi: 10.3390/sports10090126. PMID 36136381
- [Background] Phillips E, Portus M, Davids K, Renshaw I. Performance accuracy and functional variability in elite and developing fast bowlers. J Sci Med Sport. 2012 Mar;15(2):182-8. doi: 10.1016/j.jsams.2011.07.006. Epub 2011 Sep 9. PMID 21907618
- [Background] Feros SA, Young WB, O'Brien BJ. The Reliability and Sensitivity of Performance Measures in a Novel Pace-Bowling Test. Int J Sports Physiol Perform. 2018 Feb 1;13(2):151-155. doi: 10.1123/ijspp.2017-0140. Epub 2018 Feb 12. PMID 28530507
- [Background] Maker R, Taliep MS. The effects of a four weeks combined resistance training programme on cricket bowling velocity. S Afr J Sports Med. 2021 Jun 10;33(1):v33i1a9002. doi: 10.17159/2078-516X/2021/v33i1a9002. eCollection 2021. PMID 36816886
- [Background] Callaghan SJ, Govus AD, Lockie RG, Middleton KJ, Nimphius S. Not as simple as it seems: Front foot contact kinetics, muscle function and ball release speed in cricket pace bowlers. J Sports Sci. 2021 Aug;39(16):1807-1815. doi: 10.1080/02640414.2021.1898192. Epub 2021 Mar 9. PMID 33687302
- [Background] Ali K, Gupta S, Hussain ME, Alzhrani M, Manzar MD, Khan M, Alghadir AH. Effect of plyometric versus complex training on core strength, lower limb, and upper limb power in male cricketers: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2023 Nov 27;15(1):160. doi: 10.1186/s13102-023-00771-8. PMID 38008712
- [Background] Boudreau SL, Mattes LL, Lowenstein NA, Matzkin EG, Wilcox RB 3rd. Customizing Functional Rehabilitation and Return to Sport in the Female Overhead Athlete. Arthrosc Sports Med Rehabil. 2022 Jan 28;4(1):e271-e285. doi: 10.1016/j.asmr.2021.09.041. eCollection 2022 Jan. PMID 35141561